CLINICAL TRIAL: NCT07276360
Title: Phase II Randomized Non-Inferiority Trial of Hypofractionated Radiotherapy for Locally Advanced Cervical Cancer in Uganda
Brief Title: Hypofractionated Radiotherapy for the Treatment of Locally Advanced Cervical Cancer in Uganda
Acronym: HypoRTCx-UG
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uganda Cancer Institute (Other)
Collaborators: Varian Medical Systems (Industry); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U050; D43TW009759 (NIH); HS5348ES (Other: Uganda National Council for Science and Technology); Mak-SOMREC-2023-775 (Other: Makerere University School of Medicine Research Ethics Committee); RG1125359 (Other: Fred Hutch Cancer Center Institutional Review Board)
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer; Cervix Cancer; Cervical Adenocarcinoma; Cervical Small Cell Carcinoma; Cervical Adenosquamous Carcinoma
Keywords: Cervical cancer; Radiotherapy; Hypofractionation; Uganda
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiation Dose Hypofractionation; Cisplatin; Platinum; Brachytherapy; Blood Specimen Collection; Specimen Handling; Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: This is an open-label phase II randomized non-inferiority trial with a parallel group design. One hundred and twenty participants will be randomized 1:1 into two arms - conventional fractionated radiotherapy or hypofractionated radiotherapy.
Masking Description: This study does not provide for blinding of participants or providers due to the significant differences between the study intervention and control in terms of the duration of treatment, three weeks compared to five weeks of external beam radiotherapy. However, information bias will be minimized by ensuring that data collectors (research staff) are not directly involved in the delivery of treatment for study patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (HFRT) (Experimental): Patients undergo HFRT QD, Monday-Friday, for 5 fractions weekly for 16 fractions in the absence of disease progression or unacceptable toxicity. Starting on day 1 of radiation therapy, patients receive cisplatin infusion over 1 hour QW during radiation therapy. Starting by week 4, patients may also undergo HDR brachytherapy twice weekly for a total of 4 doses. Patients ineligible for brachytherapy undergo a sequential external beam boost. Additionally, patients undergo CT and blood sample collection throughout the study.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Drug: Cisplatin; Radiation: High-Dose Rate Brachytherapy; Radiation: External Beam Radiotherapy Boost; Procedure: Computed Tomography; Procedure: Biospecimen Collection; Other: Questionnaire and Physical Exam
- Arm II (CFRT) (Active Comparator): Patients undergo CFRT QD, Monday-Friday, for 5 fractions weekly for up to 25 fractions in the absence of disease progression or unacceptable toxicity. Starting on day 1 of radiation therapy, patients receive cisplatin infusion over 1 hour QW during radiation therapy. Starting by week 4, patients may also undergo HDR brachytherapy twice weekly for a total of 4 doses. Patients ineligible for brachytherapy undergo a sequential external beam boost. Additionally, patients undergo CT and blood sample collection throughout the study.
  Interventions: Radiation: Conventional Fractionated Radiotherapy; Drug: Cisplatin; Radiation: High-Dose Rate Brachytherapy; Radiation: External Beam Radiotherapy Boost; Procedure: Computed Tomography; Procedure: Biospecimen Collection; Other: Questionnaire and Physical Exam

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergoing HFRT - The prescription dose will be 40 Gy in 16 fractions (2.5 Gy/fraction) to the entire pelvis, with concurrent integrated nodal boost at 3.0 Gy per fraction (48 Gy) to involved (positive) pelvic nodes, delivered once a day, Monday through Friday, 5 fractions per week, using volumetric modulated arc therapy (VMAT).
  Other Names: Hypofractionated; hypofractionated radiotherapy; Hypofractionation; Moderately Hypofractionated Radiotherapy
  Arms: Arm I (HFRT)
Radiation: Conventional Fractionated Radiotherapy — Undergoing CFRT
  Other Names: Normofractionated Radiotherapy; Conventionally Fractionated Radiotherapy
  Arms: Arm II (CFRT)
Drug: Cisplatin — Undergoing Cisplatin
  Other Names: CDDP; Abiplatin; Platinum
Radiation: High-Dose Rate Brachytherapy — Undergoing HDR Brachytherapy
  Other Names: Brachytherapy; HDR; HDR Brachytherapy; High dose brachytherapy
Radiation: External Beam Radiotherapy Boost — Undergoing external beam radiotherapy boost
  Other Names: Boost; EBRT Boost; Boost Radiotherapy; Radiotherapy Boost
Procedure: Computed Tomography — Undergoing CT scan
  Other Names: CAT scan; CAT; Planning CT scan; CT scan; Computed Axial Tomography; Computed Axial Tomography Scan
Procedure: Biospecimen Collection — Undergoing blood sample collection
  Other Names: Blood sample; Biological sample collection; Biospecimen collected; Specimen collection
Other: Questionnaire and Physical Exam — Ancillary Studies
  Other Names: CRF; Questionnaire; Assessment; Physical Exam

SUMMARY:
This phase II trial compares the effect of hypofractionated radiotherapy (HFRT) to conventional fractionated radiotherapy (CFRT) when given in combination with cisplatin and brachytherapy in patients with stage IB3, II, or III cervical cancer. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. CFRT delivers the total dose of radiation over the amount of time according to standard practice. HFRT delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. HFRT shortens treatment duration and may reduce costs and may improve the completion rates. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Brachytherapy, also known as internal radiation therapy, uses radioactive material placed directly into or near a tumor to kill tumor cells. HFRT may be safe, tolerable, and/or as effective as CFRT when given in combination with cisplatin and brachytherapy in treating patients with stage IB3, II or III cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, and efficacy of hypofractionated radiotherapy (40 Gy in 16 fractions) compared to conventional fractionated radiotherapy (45 Gy in 25 fractions) in women with locally advanced cervical cancer in Uganda.

SPECIFIC OBJECTIVES:

I. To compare the incidence of grade 3+ gastrointestinal and genitourinary toxicity at 1- and 2-years post-treatment with hypofractionated radiotherapy (40 Gy in 16 fractions) and conventional fractionated radiotherapy (45 Gy in 25 fractions) in women with cervical cancer in Uganda.

II. To evaluate and compare local control and cervical cancer-specific survival rates at 1 and 2 year after hypofractionated radiotherapy (40 Gy in 16 fractions) versus conventional radiotherapy (45 Gy in 25 fractions).

III. To determine the association between stage-adjusted mean squamous cell carcinoma antigen (SCC-Ag) at 1-month post-treatment with the progression-free survival at 1- and 2- years post-treatment with hypofractionated radiotherapy (40 Gy in 16 fractions) or conventionally fractionated radiotherapy (45 Gy in 25 fractions).

IV. To compare the costs of healthcare to patients with cervical cancer treated with hypofractionated radiotherapy (40 Gy in 16 fractions) versus conventional fractionated radiotherapy (45 Gy in 25 fractions).

V. To evaluate patient-reported outcomes and quality of life in patients with cervical cancer treated with hypofractionated radiotherapy (40 Gy in 16 fractions) versus conventional fractionated radiotherapy (45 Gy in 25 fractions).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (INTERVENTION): Patients undergo HFRT once daily (QD), Monday-Friday, for 5 fractions weekly for 16 fractions in the absence of disease progression or unacceptable toxicity. Starting on day 1 of radiation therapy, patients receive cisplatin infusion over 1 hour once weekly (QW) during radiation therapy. Starting by week 4, patients may also undergo high dose rate (HDR) brachytherapy twice weekly for a total of 4 doses. Patients ineligible for brachytherapy undergo a sequential external beam boost. Additionally, patients undergo computed tomography (CT) and blood sample collection throughout the study.

ARM II (CONTROL): Patients undergo CFRT QD, Monday-Friday, for 5 fractions weekly for up to 25 fractions in the absence of disease progression or unacceptable toxicity. Starting on day 1 of radiation therapy, patients receive cisplatin infusion over 1 hour QW during radiation therapy. Starting by week 4, patients may also undergo HDR brachytherapy twice weekly for a total of 4 doses. Patients ineligible for brachytherapy undergo a sequential external beam boost. Additionally, patients undergo CT and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30, 90, 180, 360, 540, and 720 days.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older
* Histologically confirmed squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the uterine cervix without prior treatment
* Federation of Gynecology and Obstetrics (FIGO) 2018 stage IB3, IIA, IIB, IIIA, IIIB, or IIIC
* Able to provide written informed consent in English, Luganda, Runyankole, or Lango
* Willing to attend post-treatment follow-up for up to 12 months
* Fit for concurrent chemotherapy with cisplatin
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 2
* Absolute neutrophil count ≥ 1,500 cells/mm^3 (1.5 x 10^9/L)
* Platelets ≥ 100,000 cells/mm^3 (100 x 10^9/L)
* Hemoglobin ≥ 9.0 g/dL
* Leukocyte count ≥ 4,000 cells/mm^3 (4.0 x 10^9/L)
* Creatinine clearance > 60 mL/mins, calculated using the Cockcroft-gault equation for women
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the upper limit of normal (ULN)
* Total bilirubin < 2 x ULN unless attributed to the use of antiretroviral therapy (ART)
* HIV-positive participants must be on a stable ART regimen for at least 6 weeks prior to enrollment

Exclusion Criteria:

* Prior hysterectomy. Women with previous total or subtotal hysterectomy have no cervix, and hence the anatomical changes have an impact on the radiotherapy field, and dose prescriptions because they tend to have a higher risk for bowel toxicity from pelvic radiotherapy. Therefore, these women will be excluded due to the likely impact on the results of our study intervention
* Clinical and/or radiological evidence of distant metastases
* Prior pelvic or abdominal radiotherapy
* Presence of bilateral hip prosthesis that could interfere with radiotherapy treatment
* History of inflammatory bowel disease or any other condition that could complicate radiotherapy treatment
* Participants who are pregnant at the time of enrollment. Pregnant women have a potential risk of radiation exposure to developing fetus, which may result in fetal malformations, growth retardation, or even fatal death. Secondly, their physiological changes alter the pharmacokinetics and pharmacodynamics of concurrent chemotherapy. Therefore, to protect the health of the mother and the unborn child, pregnant women will be excluded from the study. Patients who are found to be pregnant after enrollment will have the study procedures terminated
* Concurrent untreated invasive malignancy
* Uncontrolled concurrent medical/psychiatric diagnosis that would limit compliance with study requirements
* Uncontrolled HIV infection, especially HIV viral load > 2,000 copies/mL
* Participants with CD4 counts < 200 cells/mm^3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 90 days post-treatment
  It will be categorized into 5 grades. The Conchran-Mantel-Haenszel test will be used to compare differences in the grades of AEs between patients who will receive hypofractionated radiotherapy versus conventional fractionated radiotherapy by stratifying for HIV status. A p-value of < 5% will be regarded as significant.
Incidence of grade 3 or greater radiotherapy-related gastrointestinal or genitourinary AEs | At 1 and 2 years post-treatment
  Will compare the proportion of patients between the hypofractionated radiotherapy and conventional fractionated radiotherapy using a risk difference approach, and the 95% confidence interval (CI) for the difference in proportion will be estimated using the Farrington-Manning test. Non-inferiority will be determined when the upper bound of a two-sided 95% CI is less than 10%.
Local control (complete remission, stable disease, and partial response) rate | At 1 and 2 years post-treatment
  Will be compared using means, medians, standard deviations, and ranges for continuous variables and frequencies and percentages for categorical variables. Differences in local control for each treatment group and the 95% CI will be calculated using the Chi-square test or Fisher's exact test. Data on tumor sizes that are normally distributed will be presented as means and standard deviations with 95% CI. The log-rank test will be used to compare the local control rates. The mean difference between groups will be calculated using an independent T-test for normally distributed data. Will compare the proportion between arms using a risk difference approach and the 95% CI, the difference in proportion will be estimated using the Farrington-Manning test. Non-inferiority will be determined when the upper bound of a two-sided 95% Confidence interval is less than 10%.

SECONDARY OUTCOMES:
Cervical cancer-specific survival | At 1 and 2 years post-treatment
  Will be estimated for both groups using the Kaplan-Meier method. Non-inferiority will be declared when the upper bound of the two-sided 95% CI hazard ratio is less than 1.1. Multivariable Regression analysis will be used to estimate the association between the treatment arm and local control while adjusting for potential confounders such as age, stage, and hemoglobin level.
Progression-free survival (PFS) | From randomization to the date of first recurrence or progression of disease or death, assessed up to 2 years
  Will be computed using the Kaplan-Meier survival curves, describing the median PFS and its 95% CI.

OTHER OUTCOMES:
Squamous cell carcinoma antigen (SCC-Ag) | At baseline, at 4 weeks post-treatment
  It will be assessed using an enzyme-linked immunosorbent assay. A "positive biochemical response" is defined as a decrease in SCC-Ag levels after treatment, whereas a "negative biochemical response" is defined as an increase in SCC-Ag levels after treatment based on an increase in SCC-Ag values exceeding 1 ng/mL. Will be presented as means, medians, standard deviations, and ranges. Differences in SCC-Ag levels at the end of treatment between groups and the 95% CI will be calculated. A multivariable linear regression model will be used to adjust SCC-Ag levels for the cancer stage.
Association of SCC-Ag levels and PFS | Up to 1 and 2 years post-treatment
  The Pearson or Spearman correlation coefficients will be used to estimate the association between stage-adjusted SCC-Ag levels and PFS. Cox proportional hazards regression models will be used to determine the correlation between stage-adjusted SCC-Ag levels and PFS.
Health-related quality of life (costs of healthcare) | Up to 2 years post-treatment
  The total cost per patient, the differences between the costs in the two arms, and the 95% CI will be calculated. The volume of resources and costs will mainly be reported as mean values with standard deviations and mean differences with 95% CI using an independent student t-test. All analysis will be conducted using Stata version 16.0.
Patient-reported outcomes and quality of life | Up to 2 years post-treatment
  Will be calculated, and reported in mean scores, with standard deviation and/or 95% CI. The mean score will be compared between arms with Welch's t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Solomon Kibudde, MBChB, MMed., Principal Investigator — Uganda Cancer Institute
Locations (1):
- Uganda Cancer Institute, Kampala, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No